CLINICAL TRIAL: NCT04621136
Title: PhaseI/II Investigator-Initiated Trial to Investigate Safety and Efficacy of Ripasudil in Patients With Retinopathy of Prematurity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyushu University (Other)
Responsible Party: Principal Investigator, Mitsuru Arima, Center for Clinical and Translational Research, Kyushu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTR180-01
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; ROP
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ripasudil eye drops (Experimental): Ripasudil eye drops
  Interventions: Drug: Ripasudil ophthalmic solution 0.4%

INTERVENTIONS:
Drug: Ripasudil ophthalmic solution 0.4% — Phase1 A total of three infants will receive ripasudil eye drops(0.4%) once daily for one week, followed by twice-daily drug administration for two weeks. The three infants who participate in Phase1 can continue to receive the eye drop treatment for additional 9 weeks(12 weeks in total)if the investigators determine that there are no safety issues with ripasudil. In addition, a data and safety monitoring board(DSMB)will be held two times to decide whether the new patients can be enrolled into phase1, and also if phase2 can begin.
  Phase2:A total of 21 patients will receive ripasudil eye drops(0.4%)twice daily for 12 weeks.
  Other Names: GLANATEC ophthalmic solution 0.4%

SUMMARY:
This is an open-label, single-arm phase I/II trial to evaluate the safety and efficacy of Rho-associated protein kinase(ROCK) inhibitor Ripasudil eye drops for preterm infants with Retinopathy of Prematurity(ROP).

DETAILED DESCRIPTION:
Ripasudil eye drops will be administrated to all enrolled preterm infants with zone I/II stage 1 or greater ROP （except for aggressive posterior ROP, Type1 ROP ）.

The safety and efficacy of ripasudil in treated patients will be assessed in comparison to a historical control.

ELIGIBILITY:
Inclusion Criteria:

* 1. Informed consent signed by parents or legal guardians of the patient
* 2. Patients born with less than or equal to 32 weeks of gestational age and/or less than or equal to 1,500 grams of birth weight
* 3. Patients with the following types of ROP in both eyes

  1. Zone I ROP with stage greater than or equal to 1
  2. Zone II ROP with stage greater than or equal to 1

Exclusion Criteria:

* 1. Patients with aggressive posterior ROP in one or both eyes
* 2. Patients with type 1 ROP in one or both eyes
* 3. Patients with a confirmed or suspected chromosomal abnormality or genetic disorder
* 4. History of hypersensitivity to ripasudil (including drugs with similar chemical structure) in patients or their mothers
* 5. Patients or their mothers have participated in another intervention study and have used the study drug of another intervention study within 30 days prior to enrollment in this study or within 5 times the half-life of the study drug
* 6. Patients with an ocular structural abnormality that can affect the evaluation of this clinical study by investigators
* 7. Patients with a clinically significant neurological disease (e.g., intraventricular hemorrhage grade 3 or higher, severe hydrocephalus with significantly increased intracranial pressure)
* 8. Patients with inadequate blood access
* 9. Patients with complications, allergies, or worsening systemic conditions that make it difficult to conduct this trial
* 10. Patients judged unsuitable by investigators

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Adverse Events(AEs) and Adverse Drug Reactions(ADRs) | throughout the study duration(up to week16)
  Safety Assessment

SECONDARY OUTCOMES:
Proportion of patients whose ROP worsens to Type1 ROP in one or both eyes | week12 of treatment
  Efficacy Assessment： ripasudil-treated patients will be assessed in comparison to the medical records of a historical control group
Proportion of patients with ROP remission in both eyes | week12 of treatment
  Efficacy Assessment： ripasudil-treated patients will be assessed in comparison to the medical records of a historical control group
Concentration of ripasudil and its metabolite M1 | throughout the study duration(up to week12)
  Pharmacokinetics, the population pharmacokinetic(popPK)

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuru Arima, MD,PhD, Principal Investigator — Kyushu University Hospital
Locations (3):
- Japan (3):
  - University Hospital of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Kyushu University Hospital, Fukuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamaguchi M, Nakao S, Arita R, Kaizu Y, Arima M, Zhou Y, Kita T, Yoshida S, Kimura K, Isobe T, Kaneko Y, Sonoda KH, Ishibashi T. Vascular Normalization by ROCK Inhibitor: Therapeutic Potential of Ripasudil (K-115) Eye Drop in Retinal Angiogenesis and Hypoxia. Invest Ophthalmol Vis Sci. 2016 Apr 1;57(4):2264-76. doi: 10.1167/iovs.15-17411. PMID 27124322
- [Derived] Arima M, Inoue H, Nakao S, Misumi A, Suzuki M, Matsushita I, Araki S, Yamashiro C, Takahashi K, Ochiai M, Yoshida N, Hirose M, Kishimoto J, Todaka K, Hasegawa S, Kimura K, Kusuhara K, Kondo H, Ohga S, Sonoda KH. Study protocol for a multicentre, open-label, single-arm phase I/II trial to evaluate the safety and efficacy of ripasudil 0.4% eye drops for retinopathy of prematurity. BMJ Open. 2021 Jul 27;11(7):e047003. doi: 10.1136/bmjopen-2020-047003. PMID 34315793